CLINICAL TRIAL: NCT02718222
Title: Studying the Impact and Performance of Institutionalizing Immediate Post-partum IUD Services as a Routine Part of Antenatal Counseling and Delivery Room Services in Nepal, Sri Lanka, Tanzania
Brief Title: Impact and Performance of Institutionalizing Immediate Post-partum IUD Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: International Federation of Gynaecology and Obstetrics (Other)
Responsible Party: Principal Investigator, Iqbal Shah, Principal Research Scientist, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 6904190-01
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Contraception
Keywords: Post-partum intrauterine device (PPIUD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3-9 months PPIUD intervention (Experimental): Tanzania: Baseline (no intervention) period is 9 months. Post-partum IUD intervention begins after 9 months and continues for 3 months.
  Nepal and Sri Lanka: Baseline (no intervention) period is 9 months. Post-partum IUD intervention begins after 9 months and continues for 9 months.
  Interventions: Device: Post-partum IUD
- 9-15 months PPIUD intervention (Experimental): Tanzania: Baseline (no intervention) period is 3 months. Post-partum IUD intervention begins after 3 months and continues for 9 months.
  Nepal and Sri Lanka: Baseline (no intervention) period is 3 months. Post-partum IUD intervention begins after 3 months and continues for 15 months.
  Interventions: Device: Post-partum IUD

INTERVENTIONS:
Device: Post-partum IUD — The PPIUD intervention aims to address the postpartum contraceptive needs of women by training community midwives, health workers, doctors and delivery unit staff in postpartum IUD counselling and insertion.
  Other Names: PPIUD

SUMMARY:
Studying the impact and performance of institutionalizing immediate post-partum IUD services as a routine part of antenatal counselling and delivery room services in Sri Lanka, Tanzania, and Nepal.

DETAILED DESCRIPTION:
The International Federation of Gynaecology and Obstetrics (FIGO) has designed and is planning to implement, through its nationally-affiliated Associations of Gynaecologists and Obstetricians, an intervention program on post-partum IUD (PPIUD) services. As part of this Program, FIGO is responsible for information material, training providers, improving facilities, quality of service, and monitoring the program. Independent of the implementation, this study will measure the impact and performance of this intervention in three (Sri Lanka, Nepal and Tanzania) of the six countries participating in the FIGO project entitled: "Institutionalization of immediate post-partum IUD (PPIUD) services as a routine part of antenatal counselling and delivery room services in Sri Lanka, Kenya, India, Tanzania, Nepal and Bangladesh." The FIGO intervention will take place over a nine-month period in Tanzania (nine months in the first group of three hospitals and three months in the second group of three hospitals), and over a fifteen-month period in Nepal and Sri Lanka (fifteen months in the first group of three hospitals and nine months in the second group of three hospitals). Investigators will study both the impact of the intervention on the uptake and subsequent continued use of PPIUD and the extent to which the intervention leads to the institutionalization of postpartum IUD services in the hospitals during and after the FIGO intervention and to what extent the service diffuses to other hospitals or providers. The institutionalization and diffusion of the intervention will be measured by interviewing and following up trained providers, review of hospital records and baseline, during intervention and post-intervention facility surveys.

ELIGIBILITY:
Inclusion Criteria:

* Delivered in intervention hospital during 12-month enrollment period (Tanzania)/18-month enrollment period (Nepal and Sri Lanka)

Exclusion Criteria:

* Does not live in the country where delivered
* Tanzania only: Under age 18

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140258 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage uptake of PPIUD | Within approximately 24 hours postpartum, before discharge from the hospital.
  To ascertain what percentage of women delivering in study hospitals take uptake PPIUD, participants will be interviewed after delivery, before they are discharged from the hospital.

SECONDARY OUTCOMES:
Percentage of women receiving PPIUD counseling | Within approximately 24 hours postpartum, before discharge from the hospital.
  To ascertain what percentage of women delivering in study hospitals receive counseling on PPIUD, participants will be interviewed after delivery, before they are discharged from the hospital.
Percentage of PPIUD acceptors who have expulsions at 4-6 weeks postpartum | 6 weeks postpartum
  Participants who have not deliberately removed the PPIUD will be examined by providers at 4-6 weeks postpartum, and providers will report whether the PPIUD was expelled.
Percentage of women using modern contraception at 9 months postpartum | 9 months postpartum
  Participants will be interviewed at 9 months and asked whether they are using a modern method of contraception.
Percentage of women using modern contraception at 18 months postpartum | 18 months postpartum
  Participants will be interviewed at 18 months and asked whether they are using a modern method of contraception.
Percentage of women pregnant at 18 months postpartum | 18 months postpartum
  Participants will be interviewed at 18 months and asked whether they are pregnant.

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal H Shah, PhD, Principal Investigator — Harvard School of Public Health (HSPH); David Canning, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (3):
- Center for Research on Enviornment Health and Population Activities, Kathmandu, Nepal
- Sri Lanka College of Obstetricians and Gynecologists, Colombo, Sri Lanka
- Management and Development for Health, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Investigators intend to make a de-identified dataset available after conclusion of the study.

REFERENCES:
- [Background] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Background] Hernan MA, Brumback B, Robins JM. Marginal structural models to estimate the causal effect of zidovudine on the survival of HIV-positive men. Epidemiology. 2000 Sep;11(5):561-70. doi: 10.1097/00001648-200009000-00012. PMID 10955409
- [Background] Gong Q, Schaubel DE. Partly conditional estimation of the effect of a time-dependent factor in the presence of dependent censoring. Biometrics. 2013 Jun;69(2):338-47. doi: 10.1111/biom.12023. Epub 2013 May 2. PMID 23635094
- [Background] Eroglu K, Akkuzu G, Vural G, Dilbaz B, Akin A, Taskin L, Haberal A. Comparison of efficacy and complications of IUD insertion in immediate postplacental/early postpartum period with interval period: 1 year follow-up. Contraception. 2006 Nov;74(5):376-81. doi: 10.1016/j.contraception.2006.07.003. Epub 2006 Sep 15. PMID 17046378
- [Background] Govindarajulu US, Spiegelman D, Thurston SW, Ganguli B, Eisen EA. Comparing smoothing techniques in Cox models for exposure-response relationships. Stat Med. 2007 Sep 10;26(20):3735-52. doi: 10.1002/sim.2848. PMID 17538974
- [Background] Ross John A. and Winfrey William L. Contraceptive use, intention to use and unmet need during the extended postpartum period. International Family Planning Perspectives, 2001, 27(1): 20-27.
- [Background] Rotnitzky A, Robins JM. Semiparametric regression estimation in the presence of dependent censoring. Biometrika. 1995 Dec;82(4):805-20.
- [Background] Winfrey, William and Rakesh Kshitiz. Use of Family Planning in Postpartum Period. DHS Comparative Report No. 36. 2014. Rockville, Maryland, USA: ICF International.
- [Background] Medical Eligibility Criteria for Contraceptive Use: A WHO Family Planning Cornerstone. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138639/ PMID 23741782
- [Background] Chen BA, Reeves MF, Hayes JL, Hohmann HL, Perriera LK, Creinin MD. Postplacental or delayed insertion of the levonorgestrel intrauterine device after vaginal delivery: a randomized controlled trial. Obstet Gynecol. 2010 Nov;116(5):1079-87. doi: 10.1097/AOG.0b013e3181f73fac. PMID 20966692
- [Background] Kapp N, Curtis KM. Intrauterine device insertion during the postpartum period: a systematic review. Contraception. 2009 Oct;80(4):327-36. doi: 10.1016/j.contraception.2009.03.024. Epub 2009 Aug 29. PMID 19751855
- [Background] Grimes DA, Lopez LM, Schulz KF, Stanwood NL. Immediate postabortal insertion of intrauterine devices. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD001777. doi: 10.1002/14651858.CD001777.pub3. PMID 20556754
- [Background] McKaig, Catherine and Blanchard, Holly. The IUD: A contraceptive option for postpartum and postabortion women. Access/USAID.
- [Background] Mohamed SA, Kamel MA, Shaaban OM, Salem HT. Acceptability for the use of postpartum intrauterine contraceptive devices: Assiut experience. Med Princ Pract. 2003 Jul-Sep;12(3):170-5. doi: 10.1159/000070754. PMID 12766335
- [Background] Bryant AG, Kamanga G, Stuart GS, Haddad LB, Meguid T, Mhango C. Immediate postpartum versus 6-week postpartum intrauterine device insertion: a feasibility study of a randomized controlled trial. Afr J Reprod Health. 2013 Jun;17(2):72-9. PMID 24069753
- [Background] Arrowsmith ME, Aicken CR, Saxena S, Majeed A. Strategies for improving the acceptability and acceptance of the copper intrauterine device. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008896. doi: 10.1002/14651858.CD008896.pub2. PMID 22419340
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Pagel C, Prost A, Lewycka S, Das S, Colbourn T, Mahapatra R, Azad K, Costello A, Osrin D. Intracluster correlation coefficients and coefficients of variation for perinatal outcomes from five cluster-randomised controlled trials in low and middle-income countries: results and methodological implications. Trials. 2011 Jun 14;12:151. doi: 10.1186/1745-6215-12-151. PMID 21672223
- [Background] Ali MMS, Rachael K, Cleland John, Ngo Thoai D, and Shah Iqbal H. Long-term contraceptive protection, discontinuation and switching behaviour: intrauterine device (IUD) use dynamics in 14 developing countries. London: World Health Organization and Marie Stopes International, 2011.
- [Background] Family Health Bureau MoH, Sri Lanka. Annual Report on Family Health 2012. Colombo, Sri Lanka: Ministry of Health, Sri Lanka, 2012.
- [Background] Ministry of Health and Population (MOHP) [Nepal], New ERA, and ICF International Inc. Nepal Demographic and Health Survey 2011. Kathmandu, Nepal: Ministry of Health and Population, New ERA, and ICF International, Calverton, Maryland, 2012.
- [Derived] Pearson E, Senderowicz L, Pradhan E, Francis J, Muganyizi P, Shah I, Canning D, Karra M, Ulenga N, Barnighausen T. Effect of a postpartum family planning intervention on postpartum intrauterine device counseling and choice: evidence from a cluster-randomized trial in Tanzania. BMC Womens Health. 2020 May 12;20(1):102. doi: 10.1186/s12905-020-00956-0. PMID 32398077
- [Derived] Karra M, Pearson E, Pradhan E, de Silva R, Samarasekera A, Canning D, Shah I, Weerasekera D, Senanayake H. The effect of a postpartum IUD intervention on counseling and choice: Evidence from a cluster-randomized stepped-wedge trial in Sri Lanka. Trials. 2019 Jul 8;20(1):407. doi: 10.1186/s13063-019-3473-6. PMID 31287021
- [Derived] Pradhan E, Canning D, Shah IH, Puri M, Pearson E, Thapa K, Bajracharya L, Maharjan M, Maharjan DC, Bajracharya L, Shakya G, Chaudhary P. Integrating postpartum contraceptive counseling and IUD insertion services into maternity care in Nepal: results from stepped-wedge randomized controlled trial. Reprod Health. 2019 May 29;16(1):69. doi: 10.1186/s12978-019-0738-1. PMID 31142344
- [Derived] Pradhan E, Pearson E, Puri M, Maharjan M, Maharjan DC, Shah I. Determinants of imbalanced sex ratio at birth in Nepal: evidence from secondary analysis of a large hospital-based study and nationally-representative survey data. BMJ Open. 2019 Jan 30;9(1):e023021. doi: 10.1136/bmjopen-2018-023021. PMID 30705238
- [Derived] Canning D, Shah IH, Pearson E, Pradhan E, Karra M, Senderowicz L, Barnighausen T, Spiegelman D, Langer A. Institutionalizing postpartum intrauterine device (IUD) services in Sri Lanka, Tanzania, and Nepal: study protocol for a cluster-randomized stepped-wedge trial. BMC Pregnancy Childbirth. 2016 Nov 21;16(1):362. doi: 10.1186/s12884-016-1160-0. PMID 27871269